CLINICAL TRIAL: NCT04158765
Title: Investigating the Impact of Lifestyle on Telomere Length and Telomerase Activity on Sperm Cells Originating From Infertile Men Undergoing IVF Treatment
Brief Title: The Impact of Lifestyle on Sperm Telomere Length and Telomerase Activity in Men Undergoing IVF Treatments
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0120-18-HYMC
Record Dates: First submitted 2019-07-23; First posted 2019-11-12 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen sperm and whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infertile men: Men with altered spermograms (isolated teratozoospermia or oligo-astheno-teratozoospermia)
  Interventions: Other: DNeasy Tissue Kit (QIAGEN Inc., Mississauga, Ontario, Canada) and PCR- based assay (TRAPeze Telomerase Detection Kit; Millipore, Billerica, MA).

INTERVENTIONS:
Other: DNeasy Tissue Kit (QIAGEN Inc., Mississauga, Ontario, Canada) and PCR- based assay (TRAPeze Telomerase Detection Kit; Millipore, Billerica, MA). — DNA will be extracted from sperm using the DNeasy Tissue Kit and Telomerase activity in samples will be measured using a PCR- based assay.

SUMMARY:
This aim of this study is to determine the impact of lifestyle on telomere length and telomerase enzyme activity on sperm cells of men undergoing IVF treatments.

DETAILED DESCRIPTION:
Following approval of the study by the Hospital Ethical Committee (Helsinki), semen samples and blood will be collected from infertile individuals referred to our IVF unit at Hillel Yaffe Medical Center. Informed written consent will be obtained from each participant. Standard semen analysis will be carried out according to World Health Organization protocol. An aliquot of semen sample will be used for assessment of sperm motility, concentration, and morphology by using computer-aided sperm analysis (CASA) and the remaining sample will be used for assessment of sperm telomere lengths and telomerase activity. Genomic DNA will be extracted from the remaining washed sperm and peripheral blood. Sperm telomere length will be determined by real-time polymerase chain reaction (qRT-PCR) and telomerase activity will be determined by TRAP assay (Telomeric Repeat Amplification Protocol).

ELIGIBILITY:
Inclusion Criteria:

* Infertile couple

Exclusion Criteria:

* Chronic disease
* Azoospermia

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Infertile men attending a university-affiliated IVF Unit at Hillel Yaffe Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Telomere length | Two years
  After laboratory determination of telomere length, results will be compared to lifestyle of subject to see whether smoking or other lifestyle behaviors have an effect

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Limonad, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No